CLINICAL TRIAL: NCT01507818
Title: Impact of Non-thermal Pulsed Radio Frequency (PRF)on Narcotic Use, Pain, and Health-related Quality of Life Following Shoulder Arthroscopic Rotator Cuff Repair: A Double-Blind, Randomized Sham-Controlled Trial
Brief Title: Effectiveness of the Ivivi Torino II, Pulsed Radio Frequency Device, on Narcotic Use, Pain and Quality of Life Following Shoulder Arthroscopic Rotator Cuff Repair.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amp Orthopedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Amp-PostOpShoulder-Pain-001
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Rotator Cuff Tear
Keywords: Arthroscopic Rotator Cuff Repair; Electromagnetic field treatment; Pulsed Radio Frequency treatment; Non-invasive; Non-thermal
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivivi Torino II (Active Comparator): Active treatment with Non-thermal Pulsed Radio Frequency device
  Interventions: Device: Ivivi Torino II
- Inactive Sham (Sham Comparator): Sham treatment
  Interventions: Device: Inactive Sham device

INTERVENTIONS:
Device: Ivivi Torino II — Emits a PRF generated specific electromagnetic signal consisting of a 27.12 MHz radio frequency carrier pulse-modulated with a burst duration of 3 milliseconds repeating at 2 times per second (2Hza0>
  Arms: Ivivi Torino II
Device: Inactive Sham device — The inactive control device (Sham) identical to the Active device with the exception that a PRF signal is not delivered.
  Arms: Inactive Sham

SUMMARY:
To determine the effectiveness of non-thermal PRF delivered with the Ivivi Torino II on narcotic use, pain, and health-related quality of life following shoulder arthroscopic rotator cuff surgery comparing: Active treatment versus placebo (Sham).

ELIGIBILITY:
Inclusion Criteria:

* MRI diagnosis of rotator cuff tear
* Persistent symptoms despite a minimum of 6 months of failed non-operative management
* Scheduled for primary or revision arthroscopic rotator cuff repair (with or without any of the following: debridement, subacromial decompression, distal clavicle resection, treatment of biceps tendon and /or glenoid labrum pathology, release of capsule).
* Age 40 to 80 years
* Able to read and complete English-language surveys
* Ability of the participant to comprehend the full nature and purpose of the study including possible risks and side effects
* Willingness and ability to comply with study product and methods

Exclusion Criteria:

* Diagnosis of adhesive capsulitis requiring global capsular release, instability, fracture, or arthritis
* Any implanted metallic leads, wires, or systems (e.g. pacemaker, implantable cardioverter-defibrillator)
* Known narcotic allergy, hepatitis, nephritis, or gastrointestinal ulcer
* Chronic narcotic pain medication dependency
* Vulnerable populations including prisoners, pregnant women, nursing home residents, the Investigator's students and employees, employees of sponsor, those unable to consent for themselves, uninsured subjects or others who could be subject coercion
* Worker's compensation claimant
* Medical condition, in the judgement of the patient's physician, which may interfere with the shoulder surgery or the effectiveness or safety of the study treatment
* Use of oral prednisone in the past 30 days
* Use of any investigational drug or participation in another research study within the past 30 days
* Self-reported diagnosis of autoimmune or inflammatory arthritis (e.g. Rheumatoid Arthritis, Lupus, ets.)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Average daily narcotic consumption (oxycodone mg) | week-1 post surgery
  Average, daily, patient-reported narcotic consumption (converted to oxycodone equivalents in mg) during Week 1.

SECONDARY OUTCOMES:
Average daily narcotic consumption (oxycodone mg) | Weeks 2-6 post surgery
  Average, daily, patient-reported narcotic consumption during Weeks 2-6
Visual Analogue Scale (VAS) pain | Weeks 2-6 post surgery
  Daily VAS pain (daily "current" and "maximum") during Week 1, VAS pain (daily "current" and "maximum") during Weeks 2-6
Patient-reported general health-related quality of life score (EQ-5D) | On the last day of Weeks 1-6
  The EQ-5D will be completed by the subject on the last day of each week (Weeks 1-6)
Adverse Events | Weeks 1-6 post surgery
  Adverse events will be recorded daily following randomization and analyzed for confirmation of device safety

CONTACTS AND LOCATIONS:
Overall Officials: Felix Savoie, M.D., Principal Investigator — Tulane University Schol of Medicine
Locations (3):
- United States (3):
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Mississippi sports Medicine and Orthopaedic Center, Jackson, Mississippi
  - Taos Orthopaedic Institue, Taos, New Mexico